CLINICAL TRIAL: NCT03957044
Title: The Effect of Vestibular Rehabilitation on Sensory Profile and Postrotary Nystagmus in Autistic Children
Brief Title: the Effect of Vestibular Rehabilitation in Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Physiotherapist, PhD, Associate Professor, Istinye University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Autistic Spectrum Disorder; Vestibular Disorder; Sensory Integration Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sensory integration group (Experimental): This group was given the education of sensory integration with vestibular education.
  Interventions: Other: The education of sensory integration with vestibular education
- Control group (No Intervention): The control group was given the education of sensory integration without vestibular education.

INTERVENTIONS:
Other: The education of sensory integration with vestibular education — Tactical, proprioceptive, visual and auditory senses were used in sensory integrity training sessions. In this group, the training program on tactile, proprioceptive, visual and auditory sensory activities was carried out for 2 weeks and 40 minutes. Sensory integrity training was performed by the physiotherapist and in the sensory room.
  At the end of the training sessions, mothers were informed about the application of sensory integrity training to daily activities.Sensory integrity therapy room added tactile, proprioceptive, visual and auditory sensory materials as well as materials for vestibular sensation. Vestibular sensory materials, skateboard, swing, hammock, bowl, ball, ball pool, slide, climbing bar, trampoline, and balance board were used.
  Arms: sensory integration group

SUMMARY:
This study was conducted to clarify the effect of vestibular education for autistic children on "sensory profile" and "postrotary nystagmus". In the study, the results of the two groups were compared through the treatment of sensory integration: the once who got the education and the once who did not. For this study, 26 autistic children were included who joined the " Çatalca District Unit of Disabled the Project of No Disabilities ", who was diagnosed with autism, who was 3-10 years (older than 36 months younger than 11 years). For each child, the analysis of the sensory integration and nystagmus was applied twice; at the beginning and at the end of the research. At the beginning of the research, the children were divided into two groups randomly drawn by lots. The first group was given the education of sensory integration with vestibular education and the second group was given the education of sensory integration without vestibular education. Both groups were educated for 10 weeks, 2 days a week with 40- minute sessions.

ELIGIBILITY:
Inclusion Criteria:

* The study included autistic children aged between 3 and 10 years (36 months, 11 years old) who were diagnosed with autism according to the Diagnostic and Statistical Manual of Mental Disorders criteria. The families of all children who participated in the study were informed and their written permissions were obtained.

Exclusion Criteria:

* Children who were not diagnosed with autism and who had previously received treatment for sensory integrity were excluded. The children who participated in the study had independent walking problems, those with lack of extremity, those with hip dislocation, those with postural anomalies, those who had an operation, those with infectious diseases, those with additional diagnoses with autism (such as cerebral palsy), patients with seizures, traumatic postpartum trauma, and motor development disorder. those with the postural disorder were not included in the study

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-07-01 (Actual)

PRIMARY OUTCOMES:
sensory profile test | 10 weeks
  sensory profile test
postrotary nystagmus test | 10 weeks
  postrotary nystagmus test

IPD SHARING:
Plan to Share IPD: No